CLINICAL TRIAL: NCT05733286
Title: Efficacy of Suvorexant to Improve Postoperative Sleep and Reduce Delirium Severity in Older Surgical Patients: A Double-blinded, Randomized, Placebo-controlled Trial
Brief Title: REPOSE Study: Reducing Delirium by Enhancing Postoperative Sleep With Suvorexant
Acronym: REPOSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00111869
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Delirium in Old Age
Keywords: Sleep
MeSH Terms: interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Dosing labels will be attached to each study drug dose and include pre-printed fields with
  * Protocol number
  * Personal ID number
  * Participant initials
  * Date
  * Time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suvorexant Arm (Active Comparator)
  Interventions: Drug: Suvorexant 20 mg
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant 20 mg — Administer Suvorexant versus placebo every evening for Post-Operative Day (POD) 0,1, &2
  Arms: Suvorexant Arm
Drug: Placebo — Administer Suvorexant versus placebo every evening for Post-Operative Day (POD) 0,1, &2
  Arms: Placebo Arm

SUMMARY:
This research study will evaluate the effectiveness of postoperative administration of a drug called suvorexant, to improve postoperative sleep and decrease the severity of delirium (serious confusion) in adults 65 years and older undergoing non-cardiac surgery.

DETAILED DESCRIPTION:
Suvorexant is an FDA-approved drug to treat a condition called insomnia, a sleep disorder characterized by difficulty falling asleep, staying asleep or getting good quality sleep, and has been found to have a good safety profile in older adults. Since older surgical patients often have difficulties with sleep, suvorexant might improve sleep after surgery but this remains unknown. Because difficulties with sleeping after surgery have been associated with a disorder of severe confusion called delirium, administration of suvorexant after surgery may also help prevent delirium or decrease its severity.

Participants will receive either a placebo or suvorexant by mouth (or feeding tube if present) on the first three nights after surgery while in the hospital. Prior to surgery, participants will be asked to wear a wristband sleep monitor and complete several questionnaires about their sleep, brief thinking and memory tests, a test of attention, and a measurement of their pupil size with a special camera. After surgery, participants will wear a comfortable headband device that records the electrical signals from the brain to measure the amount and depth of their sleep. This device will be worn for the first 3 nights from 9:00 PM to 6:00 AM after surgery or until hospital discharge, whichever occurs first. After surgery, participants will also answer several questions about their sleep quality and redo some of the brief thinking and memory tests (delirium tests), attention tests, and pupil size measurements. Additionally, the investigators will collect a blood sample prior to surgery and on the first two days after surgery.

Benefits of this study include the possibility of improved sleep after surgery and fewer problems with confusion and thinking and memory problems after surgery.

Risks of participation include headache, diarrhea, dry mouth, cough, abnormal dreams, dizziness, daytime tiredness and discomfort from the blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 and older
2. Undergoing non-cardiac, non-intracranial surgery, any surgical procedure not involving the skull, brain, cerebrovascular structures
3. Scheduled postoperative inpatient overnight stay
4. Able to give informed consent or has legally authorized representative able to give informed consent on their behalf
5. English-speaking

Exclusion Criteria:

1. Inmate of correctional facility
2. Body mass index> 40
3. Legal blindness
4. Unable to perform study related questionnaires and assessments
5. Use of outpatient sedating sleep aids > 2 times per any week in 1 month preceding day of surgery. Sedating sleep aids, *See list Below.
6. History of psychotic disorder, including schizophrenia, schizoaffective disorder, schizophreniform or brief psychotic disorder.
7. History of liver failure with documented international normalized ratio (INR) of >1.2 or with history of hepatic encephalopathy
8. History of severe sleep apnea or obesity hypoventilation syndrome requiring home bilevel positive airway pressure therapy or home ventilator or other forms of noninvasive ventilation
9. Chronic lung disease requiring home oxygen therapy
10. History of narcolepsy
11. Use of systemic (oral, intravenous, intramuscular, subcutaneous) moderate or strong CYP3A inhibitors within 1 week prior to surgery, *See list below
12. Use of systemic (oral, intravenous, intramuscular, subcutaneous) moderate or strong CYP3A inducers within 1 week prior to surgery, *See list below.
13. Current or planned administration of digoxin, or is currently experiencing digoxin toxicity
14. Undergoing surgery that will result in inability to take medications by mouth including laryngectomy, tracheostomy, and oral resection/reconstructive surgery
15. Undergoing surgery that will require postoperative strict bowel rest, including gastrectomy, esophagectomy, and pancreaticoduodenectomy
16. Undergoing surgery in an area that will make it unsafe to wear a headband, such as scalp or forehead procedures.
17. Inappropriate for study inclusion based on the judgement of the principal investigator

Exclusionary Medications:

Moderate CYP3A inhibitors: Amprenavir, Aprepitant, Atazanavir, Ciprofloxacin, Diltiazem, Erythromycin, Fluconazole, Fosamprenavir, Imatinib, Verapamil, grapefruit juice.

Strong CYP3A inhibitors: Ketoconazole, Itraconazole, Posaconazole, Clarithromycin, Nefazodone, Ritonavir, Saquinavir, Nelfinavir, Indinavir, Boceprevir, Telaprevir, Telithromycin, Conivaptan

Moderate/Strong CYP3A inducers: Apalutamide, Carbamazepine, Enzalutamide, Ivosidenib, lumacaftor, Mitotane, Phenytoin, Rifampin, St. John's wort, Bosentan, Cenobamate, Dabrafenib, Efavirenz, Etravirine, Lorlatinib, Pexidartinib, Phenobarbital, Primidone, Sotorasib.

Sedating sleep aids: Mirtazapine, Trazodone, Flurazepam, Temazepam, Triazolam, Estazolam, Quazepam, Clonazepam, Lorazepam, Midazolam, Alprazolam, Diazepam, Zolpidem, Zaleplon, Eszopiclone, Diphenhydramine, Doxylamine, Hydroxyzine, Suvorexant, Doxepin

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Devinney Jr, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fallon JM, Hashemaghaie M, Peterson CE, Tran D, Wu SR, Valdes JM, Pedicini NM, Adams ME, Soltis M, Mansour W, Wright MC, Raghunathan K, Treggiari MM, Sasannejad C, Devinney MJ. Protocol and design of the REPOSE study: a double-blinded, randomised, placebo-controlled trial to evaluate the efficacy of suvorexant to improve postoperative sleep and reduce delirium severity in older patients undergoing non-cardiac surgery. BMJ Open. 2025 Mar 13;15(3):e091099. doi: 10.1136/bmjopen-2024-091099. PMID 40081971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients age 65 or older scheduled for non-cardiac elective surgery with planned postoperative overnight stay at Duke University Hospital and Duke Medical Pavilion were contacted to determine interest in enrollment in this study. Patients were consented in-person at preoperative visits or via electronic consent over telephone or videoconferencing.
Pre-assignment Details: 14 participants were never assigned to a treatment arm due to screen fail (n= 4), withdrawal by PI (n = 4), subject chose to withdraw prior to surgery (n = 3), and surgery cancellation (n =3).
Groups:
- Suvorexant Arm: Administer Suvorexant every evening for Post-Operative Day (POD) 0, 1, and 2
- Placebo Arm: Administer placebo every evening for Post-Operative Day (POD) 0, 1, and 2
Period: Overall Study
Arm/Group | Suvorexant Arm | Placebo Arm
Started | 68 | 60
Completed | 66 | 57
Not Completed | 2 | 3
Not completed — Never received study drug | 2 | 3

BASELINE CHARACTERISTICS:
Population: Participants who received a dose of study drug or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant Arm | Placebo Arm | Total
Number analyzed (Participants) | 66 | 57 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (4) | 72 (5) | 72 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 38 | 34 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 57 | 46 | 103
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 62 | 54 | 116
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 57 | 123

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time (TST) on the First Postoperative Night
Description: Total sleep time (TST) on first postoperative night that patient received study drug, as measured by electroencephalography (EEG). Total sleep time includes amount of time in sleep during the lights out period (defined between 21:00 and 06:00).
Time Frame: The first postoperative night that the participants received study drug (D0)
Population: Participants with EEG data for total sleep time determination.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Suvorexant Arm | Placebo Arm
Number analyzed (Participants) | 62 | 55
hours | 3.91 (2.00) | 3.84 (2.07)
Statistical Analysis 1: Comparison: Suvorexant Arm vs Placebo Arm; Test type: Superiority; p = 0.853, t-test, 2 sided — Given an SD of approximately 35 min for TST in healthy adults, a sample size of 58 subjects per group will provide 86% power to detect a 20 min difference in TST between treatment groups using a two-sample t-test with a two-sided alpha of 0.05

2. Secondary Outcome: Peak Postoperative Delirium Severity Score
Description: Three minute Confusion Assessment Method (3D-CAM ) severity scores up through postoperative day 5 or discharge, whichever occurs first, in patients receiving suvorexant vs placebo. Scores range from 0-20 and the higher score is worse.
Time Frame: Postoperative Day 0 through Day 5
Population: Participants with 3D-CAM delirium severity scores collected.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Suvorexant Arm | Placebo Arm
Number analyzed (Participants) | 66 | 56
score on a scale | 2 [1 to 3] | 1 [1 to 3]
Statistical Analysis 1: Comparison: Suvorexant Arm vs Placebo Arm; Test type: Superiority; p = 0.340, Wilcoxon (Mann-Whitney) — Unadjusted. P < 0.05 is considered significant. A sample size of 58 patients per group will provide 80% power to detect a 0.95-point difference between treatment groups using a two-sided t-test with an alpha of 0.05

3. Other Pre Specified Outcome: Postoperative Average Electrographic Total Sleep Time Over the 3-night Recording Period
Description: Using the electrographic headband data, differences in postoperative sleep architecture (including stage 2 and 3 NREM sleep and REM sleep) will be compared in participants who received suvorexant compared to those who received placebo using two-sample t-tests. No multiple comparison correction for multiple sleep stages is planned because these are exploratory analyses. Average total sleep time over all nights that participants receive study drug will also be compared using two-sample t-tests.
Time Frame: Postoperative day 0-2
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Average Postoperative Richards-Campbell Subjective Sleep Quality Scores
Description: To assess subjective sleep quality, the Richards-Campbell subjective sleep quality questionnaire will be administered daily from postoperative day 1-5 or until hospital discharge, whichever occurs first. The total subjective sleep quality score will be compared between placebo and suvorexant groups using a two-sample t-test.
Time Frame: Postoperative days 1-5
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change In Pupil Diameter Fluctuations From Preoperative Baseline Through Postoperative Day 3
Description: Pupillary unrest under ambient light is an index of spontaneous pupil fluctuations that occur secondary to activity of the locus coeruleus, an important brainstem nucleus involved in maintenance of wakefulness and attentional control. Decreased wakefulness has been associated with decreased pupillary unrest at ambient light, suggesting that pupillary unrest at ambient light is a marker of sleep deprivation-related alterations in wakefulness and attention. Here, infrared pupillometry will be used to measure participant's pupil diameter fluctuations under ambient light conditions both before surgery and daily up through postoperative day 3. We will compare postoperative changes in pupillary unrest at ambient light in both suvorexant and placebo-treated using a two-sided t-test.
Time Frame: Preoperative baseline and postoperative days 1-3
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Average Response Latency on Preoperative and Postoperative Psychomotor Vigilance Testing
Description: Sleep deprivation results in decreased ability to sustain attention, which can be measured with the 5-minute psychomotor vigilance task. The psychomotor vigilance task measures simple reaction times to a visual stimulus over a minute to assess for slowed responses and lapses (i.e., failed response to visual stimuli). Response times, speed, and lapses will be compared between suvorexant and placebo-treated groups to see if postoperative nightly suvorexant has an effect on these sustained attention measures. Using the NASA PVT+ application on an Apple iPad, the psychomotor vigilance task will be collected before surgery, and daily on postoperative day 1-3, or until hospital discharge, whichever occurs first. Analyses will examine pre-to-postoperative change in sustained attention measures to adjust for preoperative performance variability between participants.
Time Frame: Preoperative baseline, and postoperative days 1-3
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Postoperative Hospital Length of Stay
Description: Postoperative delirium occurs in up to 40% of older surgical patients and has been associated with prolonged hospital stays, long-term cognitive impairment, and increased one-year postoperative mortality. We will record the length of hospital stay for each participant.
Time Frame: From Postoperative day 0 up to 4 week follow up visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Surgery (day 0) to 4-week follow-up call
Arm/Group | Suvorexant Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 1/66 | 0/57
Serious Adverse Events (participants affected / at risk) | 9/66 | 9/57
Other Adverse Events (participants affected / at risk) | 14/66 | 13/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant Arm (N=66) | Placebo Arm (N=57)
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Intraoperative cardiac arrest (Cardiac disorders) | 0 | 0
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 | 0
Erythematous rash (Infections and infestations) | 0 | 1
Postoperative Spinal Abscess (Infections and infestations) | 1 | 0
Postoperative Seroma Infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound dehiscence (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
Abdominal Fluid Collection (Injury, poisoning and procedural complications) | 1 | 0
acute blood loss anemia from intraoperative aortic injury (Injury, poisoning and procedural complications) | 0 | 0
Increased Postoperative Pain (Injury, poisoning and procedural complications) | 1 | 0
Surgical Incision Swelling (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1
Death due to persistent comatose state (Nervous system disorders) | 1 | 0
Intraparenchymal hemorrhage (Nervous system disorders) | 1 | 0
Multifocal Acute Brain Infarcts (Nervous system disorders) | 0 | 0
Transient Ischemic Attack (Nervous system disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Postoperative Urinoma (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemorrhagic Shock (Vascular disorders) | 0 | 0
Hypotension (Vascular disorders) | 0 | 2
Pulmonary embolism (Vascular disorders) | 1 | 0
Pulmonary Embolus (Vascular disorders) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Suvorexant Arm (N=66) | Placebo Arm (N=57)
Leg Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Self-reported somnolence (Nervous system disorders) | 2 | 1
Observed somnolence (Nervous system disorders) | 8 | 7
Abnormal Dreams (Psychiatric disorders) | 3 | 5
Hypnagogic Hallucinations (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT05733286/Prot_SAP_000.pdf